CLINICAL TRIAL: NCT06781099
Title: Feasibility, Tolerability and Efficacy of Extracorporeal Iron Purification in Patients With Myelodysplastic Syndrome or Myelofibrosis Intolerant of or Contraindicated to Oral or Subcutaneous Chelation Treatment.
Brief Title: Feasibility Trial of Extracorporeal Iron Purification in Patients With Myelodysplastic Syndrome or Myelofibrosis
Acronym: MEXIRON
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Collaborators: MEXBrain 13 avenue Albert Einstein 69100 Villeurbanne (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL23_0102; 2024-A02473-44 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2025-01-08; First posted 2025-01-17 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Myelodysplastic Syndrome; Myelofibrosis
Keywords: Myelodysplastic syndrome; myelofibrosis; iron chelation therapy; haemodialysis
MeSH Terms: conditions — Myelodysplastic Syndromes; Primary Myelofibrosis

STUDY DESIGN:
Intervention Model Description: Feasibility, prospective, monocentric, pilot clinical investigation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: low-volume continuous veno-venous haemodialysis with MEX-CD1 use (Experimental): Patients enrolled will benefit 3 consecutive cycle of low volume continuous veno-venous haemodialysis using MEX-CD1 treatment.
  Interventions: Device: Low-volume continuous veno-venous haemodialysis with MEX-CD1 use

INTERVENTIONS:
Device: Low-volume continuous veno-venous haemodialysis with MEX-CD1 use — MEX-CD1 is a hyper-chelating colloidal solution that can be added to the dialysate to be used in low-volume continuous veno-venous hemodialysis. Intervention includes 3 low-volume continuous veno-venous hemodialysis for a duration of 4 hours each. For non-hospitalized patients, the treatment is performed on an outpatient basis.

SUMMARY:
In transfusion-dependent myelodysplastic syndromes patients, regular blood transfusions lead to iron overload, which can cause organ damage, hormonal imbalances, and increased infection risk, ultimately impacting patient survival. Standard oral iron chelation therapies can be intolerable for some patients due to adverse effects. The MEX-CD1 device (class III) could potentially offer an alternative for these patients by reducing serum iron levels through a novel, extracorporeal approach.

MEXIRON clinical investigation focuses on the use of MEX-CD1, a medical device designed for extracorporeal chelation therapy to reduce serum iron overload in patients suffering from transfusion-dependent myelodysplastic syndromes (MDS) and myelofibrosis.

MEXIRON aims to evaluate the device's use feasibility, safety, and effectiveness in reducing serum free iron levels. Transfusions needs, patient experience and quality of life are also assessed.

Each enrolled patients will undergo three low-volume continuous veno-venous haemodialysis cycles within one week.

Following the three- haemodialysis cycles, patients will be monitored through on-site follow-up visits at 7 days, 28 days, and 90 days post-treatment to assess long-term effects.

ELIGIBILITY:
Inclusion Criteria:

* Patient followed for myelodysplastic syndrome or myelofibrosis.
* Patient with platelet count ≥50 giga/L at inclusion.
* Patients with severe anemia and hemoglobin <70 g/L at baseline.
* Patient with intolerance or contraindication to oral or subcutaneous chelation therapy.
* Ferritinemia >1000 µg/L or hepatic iron concentration ≥7 mg/g or cardiac T2* <20 ms at inclusion.
* Patient able to understand (French-speaking) and comply with protocol, having signed informed consent.

Exclusion Criteria:

* Patients with primary hemochromatosis (transferrin saturation coefficient CS-Tf > 45%).
* Patients with a contraindication to the use of MEX-CD1: weight < 30 kg, iron deficiency.
* Patients with a known allergy or contraindication to heparin or citrate.
* Patients undergoing azacitidine or other chemotherapy (or considered as such) for myelodysplastic syndrome or myelofibrosis.
* Patients with indications for allogeneic bone marrow transplantation.
* Patients with a known allergy to shellfish (MEX-CD1 contains chitosan of animal origin) or to one of the other components of MEX-CD1.
* Patients with a peripheral vascular access that is difficult to access or that needs to be preserved.
* Patients participating in other interventional research that could interfere with the results of the study.
* Patients under legal protection or unable to express their consent.
* Patients under psychiatric care.
* Patient deprived of liberty by judicial or administrative decision.
* Pregnant or breast-feeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2026-01-06 (Actual); Primary Completion 2027-01-06 (Estimated); Study Completion 2027-05-06 (Estimated)

PRIMARY OUTCOMES:
Performance of MEX-CD1 on total iron chelation during a session epuration. | Day 4
  Quantity of serum iron values measured in the dialysate bag (H0), in the effluent line (H1, H2, H3, H4), and in the effluent bag (H4) during each low-volume continuous veno-venous hemodialysis cycle

SECONDARY OUTCOMES:
Performance of MEX-CD1 on iron profile. | Day 4
  Variations in serum iron, ferritin and transferrin values from the start until i) each low-volume continuous veno-venous hemodialysis cycle ending (H4) and ii) after 3 low-volume continuous veno-venous hemodialysis cycles
Safety of MEX-CD1 use | week 16
  Assessment of adverse events during low-volume continuous veno-venous hemodialysis cycles and all follow up period.
Impact on blood products patient's needs. | week 16
  Assessment on patient's red blood cells administration from the start of the first MEX-CD1 treatment until the follow-up ending.
Feasibility of MEX-CD1 use | Day 4
  Assessment of patient's proportion who will have performed i) the entire first low-volume continuous veno-venous hemodialysis cycle and ii) the whole weakly 3 consecutive cycles at the end of the third low-volume continuous veno-venous hemodialysis cycle.
Patient's reported tolerability of low-volume continuous veno-venous hemodialysis cycle. | Day 4
  Patients tolerability assessment by Visual Analog Scales (VAS) on painful and asthenia feelings at the end of each low-volume continuous veno-venous hemodialysis cycle.
Patient's reported quality of life. | Week 16
  Quality of life assessment by the Medical Outcome Study Short Form 12 from the inclusion visit until end of follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Lyon Sud, Oullins-Pierre-Bénite, France